CLINICAL TRIAL: NCT04736940
Title: Definition of Crises in Medical Oncology: a Two-way Perspective of Patients and Caregivers, a Prospective Observational Study.
Brief Title: Definition of Crises in Medical Oncology: a Two-way Perspective of Patients and Caregivers. The COPE Study. (COPE)
Acronym: COPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Canceropôle Ile de France (Unknown)
Responsible Party: Sponsor
Other Study IDs: En attente de promotion
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Crises Situations That the Patients and Caregivers Confront in Daily Practice
Keywords: Conflict psychological; patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients: Patients followed or currently treated for a solid or haematological neoplasia
- Doctors: Medical oncologist or haematologist
- Paramedical staff: Nurses or assistant nurses
- Oncopsychologist: Psychologist specialised in the care of patients with cancer

SUMMARY:
Our objective is to identify the main crises facing the patients and caregivers in medical oncology and rank them by order of importance. Each group of participant will also express its perception of other participants' list of crises.

DETAILED DESCRIPTION:
Hypotheses:

Crises in medical oncology need to be precisely defined and classified. It should be the first step to offer appropriate support and solutions, improve communication and eventually improve quality of life/work for caregivers and for patients. Crises in medical oncology can imply all actors: doctors, nursing staff, psychologists, administration and patients. The definition of crisis and the level of importance of each situation may vary among these different groups. Nevertheless, we expect to identify shared characteristics. Patients' point of view which is rarely expressed will be collected. This work will also bring a better understanding of the perception each group have of each other.

Objectives:

Our main objective is to identify the main crises facing the patients and caregivers in medical oncology and rank them by order of importance. Each actor will also express its perception of other actors' list of crises.

Methods:

This work is led by an innovative multidisciplinary team of investigators associating patients, oncopsychologists, nurses and oncologists. Four study groups of participants are composed: a group of patients, a group of oncopsychologists, a group nurses and a group of oncologists.

Demographic characteristics, general characteristics of the disease for the patients or type of exercise for the caregivers are collected.

The first step of the project is to establish a list of crisis situations in each group consisting of 10 participants. The methodology applied is a modify Delphi in three rounds via a digital survey. In the first round, participants react to a pre-existing list, and are invited to complete it. The content is then analyzed, classified and developed into a list emailed for the second round.

In a second round, the participants establish a ranking of the items on a scale of 1-6 (not important to extremely important). The group of patients will then rank the items added by the caregivers, and vice-versa.

During the third and last round, the average of items is presented and the participants submit a new ranking. Individual interviews will be held to comment the results.

The second step of the project enables to widen the study population, with a minimal objective of 100 participants per group. These new participants receive the list established in the first step to grade 20 items per frequency and importance.

ELIGIBILITY:
Inclusion Criteria:

- For patients: History of neoplasia or active treatment for a neoplasia of any localization of any phase.

No restriction of center of treatment >18 years old Written consent must be obtained before any data collection

- For caregivers Being a doctor, nurse, or a psychooncologist No restriction of age, or seniority

Exclusion Criteria

- For patients: Patients who participate 1st step cannot participate to 2nd step

- For caregivers Caregivers who participate 1st step cannot participate to 2nd step.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from public or private clinics or hospitals involved in oncology in France Communication on the study to recruit participants is done widely via professional of patients' networks
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
List of crises ranked by order of importance in each group of paticipant | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Olivier HUILLARD, PhD, Study Chair — APHP Assistance Publique des Hôpitaux de Paris; Zahra CASTEL AJGAL, MD, Principal Investigator — APHP Assistance Publique des Hôpitaux de Paris
Locations (1):
- APHP Assistance Publique des Hôpitaux de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carnevale FA, Farrell C, Cremer R, Canoui P, Seguret S, Gaudreault J, de Berail B, Lacroix J, Leclerc F, Hubert P. Struggling to do what is right for the child: pediatric life-support decisions among physicians and nurses in France and Quebec. J Child Health Care. 2012 Jun;16(2):109-23. doi: 10.1177/1367493511420184. Epub 2012 Jan 13. PMID 22247181
- [Background] Coast J, Bailey C, Orlando R, Armour K, Perry R, Jones L, Kinghorn P. Adaptation, Acceptance and Adaptive Preferences in Health and Capability Well-Being Measurement Amongst Those Approaching End of Life. Patient. 2018 Oct;11(5):539-546. doi: 10.1007/s40271-018-0310-z. PMID 29744765
- [Background] Hong P, Maguire E, Purcell M, Ritchie KC, Chorney J. Decision-Making Quality in Parents Considering Adenotonsillectomy or Tympanostomy Tube Insertion for Their Children. JAMA Otolaryngol Head Neck Surg. 2017 Mar 1;143(3):260-266. doi: 10.1001/jamaoto.2016.3365. PMID 27930764
- [Background] Bochatay N, Bajwa NM, Cullati S, Muller-Juge V, Blondon KS, Junod Perron N, Maitre F, Chopard P, Vu NV, Kim S, Savoldelli GL, Hudelson P, Nendaz MR. A Multilevel Analysis of Professional Conflicts in Health Care Teams: Insight for Future Training. Acad Med. 2017 Nov;92(11S Association of American Medical Colleges Learn Serve Lead: Proceedings of the 56th Annual Research in Medical Education Sessions):S84-S92. doi: 10.1097/ACM.0000000000001912. PMID 29065028
- [Background] Walrath JM, Dang D, Nyberg D. An organizational assessment of disruptive clinician behavior: findings and implications. J Nurs Care Qual. 2013 Apr-Jun;28(2):110-21. doi: 10.1097/NCQ.0b013e318270d2ba. PMID 23072933
- [Background] Knickle K, McNaughton N, Downar J. Beyond winning: mediation, conflict resolution, and non-rational sources of conflict in the ICU. Crit Care. 2012 Jun 19;16(3):308. doi: 10.1186/CC11141. PMID 22713247
- [Background] Back AL, Arnold RM. Dealing with conflict in caring for the seriously ill: "it was just out of the question". JAMA. 2005 Mar 16;293(11):1374-81. doi: 10.1001/jama.293.11.1374. PMID 15769971
- [Background] Chiarchiaro J, White DB, Ernecoff NC, Buddadhumaruk P, Schuster RA, Arnold RM. Conflict Management Strategies in the ICU Differ Between Palliative Care Specialists and Intensivists. Crit Care Med. 2016 May;44(5):934-42. doi: 10.1097/CCM.0000000000001583. PMID 26765500
- [Background] Park M, Jeon SH, Hong HJ, Cho SH. A comparison of ethical issues in nursing practice across nursing units. Nurs Ethics. 2014 Aug;21(5):594-607. doi: 10.1177/0969733013513212. Epub 2014 Jan 21. PMID 24449700
- [Background] Breslin JM, MacRae SK, Bell J, Singer PA; University of Toronto Joint Centre for Bioethics Clinical Ethics Group. Top 10 health care ethics challenges facing the public: views of Toronto bioethicists. BMC Med Ethics. 2005 Jun 26;6:E5. doi: 10.1186/1472-6939-6-5. PMID 15978136
- [Background] Killen AR, Fry ST, Damrosch S. Ethics and human rights issues in perioperative nurses: a subsample of Maryland nurses. Semin Perioper Nurs. 1996 Apr;5(2):77-83. PMID 8718399
- [Background] Hsu C-C, Sandford BA. The Delphi Technique: Making Sense Of Consensus n.d.;12:8.
- [Background] Blackwood B, Albarran JW, Latour JM. Research priorities of adult intensive care nurses in 20 European countries: a Delphi study. J Adv Nurs. 2011 Mar;67(3):550-62. doi: 10.1111/j.1365-2648.2010.05512.x. Epub 2010 Nov 23. PMID 21091912
- [Background] Meskell P, Murphy K, Shaw DG, Casey D. Insights into the use and complexities of the Policy Delphi technique. Nurse Res. 2014 Jan;21(3):32-9. doi: 10.7748/nr2014.01.21.3.32.e342. PMID 24460564
- [Background] Démographie des professionnels de santé : qui sont les médecins en 2018 ? Quelle accessibilité aux médecins généralistes ? Combien d'infirmiers en 2040 ? Un outil de projections d'effectifs de médecins - Ministère des Solidarités et de la Santé n.d. http://drees.solidarites-sante.gouv.fr/etudes-et-statistiques/publications/communiques-de-presse/article/demographie-des-professionnels-de-sante-qui-sont-les-medecins-en-2018-quelle.
- [Background] La profession d'infirmière : situation démographique et trajectoires professionnelles - Data.gouv.fr n.d. /fr/datasets/la-profession-d-infirmiere-situation-demographique-et-trajectoires-professionnelles-30378340/ .